CLINICAL TRIAL: NCT05530356
Title: Renal Hemodynamics, Energetics and Insulin Resistance in Youth Onset Type 2 Diabetes: A Follow-up Study
Brief Title: Renal Hemodynamics, Energetics and Insulin Resistance: A Follow-up Study
Acronym: HEIRitage
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-2961
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes; Diabetes Type 2; Diabetic Nephropathies; Nephropathy; Obesity; Adolescent Obesity; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Kidney Diseases; Obesity; Pediatric Obesity | interventions — p-Aminohippuric Acid; Iohexol; Dextrans; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples to be retained will include urine, plasma, and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lean Controls (previously enrolled in the Renal HEIR Study)
  Interventions: Drug: Aminohippurate Sodium Inj 20%; Drug: Iohexol Inj 300 MG/ML; Drug: Dextran 40
- Obese Youth without Type 2 Diabetes (previously enrolled in the Renal HEIR Study)
  Interventions: Drug: Aminohippurate Sodium Inj 20%; Drug: Iohexol Inj 300 MG/ML; Drug: Dextran 40; Radiation: Positron Emission Tomography
- Obese Youth with Type 2 Diabetes (previously enrolled in the Renal HEIR Study)
  Interventions: Drug: Aminohippurate Sodium Inj 20%; Drug: Iohexol Inj 300 MG/ML; Drug: Dextran 40; Procedure: Renal Biopsy; Radiation: Positron Emission Tomography

INTERVENTIONS:
Drug: Aminohippurate Sodium Inj 20% — Diagnostic aid/agent used to measure effective renal plasma flow (ERPF)
  Other Names: Sodium 4-amino hippurate (PAH) inj 20% 2g/10mL; Para-aminohippurate; Aminohippuric acid
Drug: Iohexol Inj 300 MG/ML — Diagnostic aid/agent used to measure glomerular filtration rate (GFR)
  Other Names: omnipaque 300
Drug: Dextran 40 — Diagnostic aid/agent used to measure glomerular size selectivity
  Other Names: Dextran; LMD
Procedure: Renal Biopsy — Minimally invasive outpatient procedure in interventional radiology to obtain renal tissue cores.
  Other Names: Kidney Biopsy
  Groups: Obese Youth with Type 2 Diabetes (previously enrolled in the Renal HEIR Study)
Radiation: Positron Emission Tomography — Imaging study performed to study renal oxidative metabolism
  Other Names: PET Scan
  Groups: Obese Youth with Type 2 Diabetes (previously enrolled in the Renal HEIR Study); Obese Youth without Type 2 Diabetes (previously enrolled in the Renal HEIR Study)

SUMMARY:
The current protocol plans to enroll participants with youth-onset Type 2 Diabetes (T2D) as well as obese and lean controls from the Renal-HEIR - Renal Hemodynamics, Energetics and Insulin Resistance in Youth Onset Type 2 Diabetes Study (n=100) [COMIRB #16-1752] in a prospective investigation that seeks to 1) define the changes in kidney function by gold standard techniques and energetics by functional Magnetic Resonance Imaging (MRI) in adolescents with and without T2D as they transition to young adulthood; 2) quantify kidney oxidative metabolism by 11C-acetate Positron Emission Tomography (PET) in a subset of participants who are ≥18 years of age with youth-onset T2D and/or obesity; 3) determine peripheral arterial stiffness by SphygmoCor. Mechanistic insight will be provided by transcriptomic analyses of repeat biopsies 3-years after their initial biopsy for eligible participants with youth-onset T2D, as well as molecular analysis of tissue obtained from J-wire endovascular biopsies. This study will also leverage this well-characterized cohort of youths to define youth-onset T2D-related changes in brain morphology and function by structural MRI and resting-state functional MRI and through the assessment of cognitive function (fluid and crystallized intelligence) using the NIH Toolbox Cognitive Battery (NIHTB-CB), as an exploratory objective. All enrollees in Renal-HEIR have consented to be contacted for future research opportunities.

ELIGIBILITY:
Inclusion Criteria:

* Obese youth with and without Type 2 Diabetes + lean controls who were previously enrolled in the Renal HEIR Study
* Participants who will undergo a PET Scan: ≥ 18 years

Exclusion Criteria:

* Anemia
* Seafood, iodine, or penicillin allergy
* Pregnancy
* MRI Scanning contraindications (claustrophobia, implantable devices, >550 lbs)
* History of bleeding or clotting disorders, thrombocytopenia, warfarin and/or heparin use
* Taking sulfonamides, procaine, thiazolsulfone or probenecid

Ages: 12 Years to 26 Years | Sex: All
Age Groups: Child, Adult
Study Population: Population to be enrolled will be comprised of obese youth with and without T2D and lean controls who were previously enrolled in the Renal-HEIR (#16-1752) study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Effective Renal Plasma Flow (ERPF) | 4 Hours
  Measured by PAH clearance
Glomerular Filtration Rate | 4 Hours
  Measured by Iohexol Clearance
Glomerular Size Selectivity | 4 hours
  Measured by Dextran sieving
Renal Oxygen Availability | 1 hour
  Measured by functional kidney MRI
Renal Perfusion | 1 hour
  Measured by functional kidney MRI + PET Scan
11-C Acetate Tracer Uptake | 1 Hour
  Measured by PET Scan
Renal Oxidative Metabolism | 1 Hour
  Measured by PET Scan
Blood Volume Fraction | 1 Hour
  Measured by PET Scan
Glomerular Basement Membrane Width | 1 Hour
  Measured by Renal Biopsy
Mesangial Expansion | 1 Hour
  Measured by Renal Biopsy
Interstitial Fibrosis | 1 Hour
  Measured by Renal Biopsy
Renal Arteriosclerosis | 1 Hour
  Measured by Renal Biopsy
Spatial Transcriptomics | 1 Hour
  Measured by Renal Biopsy
Spatial Metabolomics | 1 Hour
  Measured by Renal Biopsy

SECONDARY OUTCOMES:
Pulse Wave Velocity between Carotid and Femoral Artery | 10 minutes
  Measured by PWV
Whole brain gray matter volume | 1 Hour
  Measured by brain MRI
Whole brain cortical thickness | 1 Hour
  Measured by brain MRI
Whole brain resting-state network connectivity | 1 Hour
  Measured by brain MRI
Age-corrected composite fluid cognition score | 1 Hour
  Measured by brain MRI

CONTACTS AND LOCATIONS:
Overall Officials: Petter Bjornstad, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided